CLINICAL TRIAL: NCT01915537
Title: A Prospective Cohort Study to Observe the Difference of Efficacy Between Infliximab With Methotrexate and Classic DMARDs in the Severe Rheumatoid Arthritis Patients With Poor Prognosis
Brief Title: Infliximab and Classic DMARDs in the Rheumatoid Arthritis Patients
Acronym: INNOVATION
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhang, Xiao, M.D. (Individual)
Collaborators: Central South University (Other); Tianjin Medical University General Hospital (Other); Xijing Hospital (Other)
Responsible Party: Sponsor-Investigator, Zhang, Xiao, M.D., Director, Zhang, Xiao, M.D.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INNOVATION
Record Dates: First submitted 2013-07-30; First posted 2013-08-05 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-07

CONDITIONS: Rheumatoid Arthritis（RA）
Keywords: poor prognosis; severe RA; infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Infliximab group (Experimental): Infliximab with MTX treatment
  Interventions: Drug: Infliximab group
- Classic DMARDs treatment group (Active Comparator): Classic DMARDs treatment（MTX 、LEF 、HCQ 、 LEF ）
  Interventions: Drug: Classic DMARDs treatment group

INTERVENTIONS:
Drug: Infliximab group — Infliximab with MTX treatment: Infliximab 3mg/kg at week 0, 2, 6 and then once every 8 weeks, MTX>7.5mg per week. To observe the results at week 14, 30, 54 and 102 after 6 times IFX treatment. It recommended that continue to receiving IFX treatment after remission for a period of time in good economic condition patients while receiving MTX with HCQ or LEF in poor economic condition patients.
  Arms: Infliximab group
Drug: Classic DMARDs treatment group — Classic DMARDs treatment: combination of 2 or 3 drugs, 2-drugs combination is MTX with LEF or Thunder God Vine, 3-drugs combination is MTX with HCQ and LEF or Thunder God Vine for total 30 weeks.
  Effective dose: MTX: 10-15mg per week; LEF: 20mg per day; HCQ: 200-400 mg per day; Thunder God Vine: 40-60 mg per day; It recommended that the maintain regimen is MTX with HCQ or LEF after remission for a period of time.
  Arms: Classic DMARDs treatment group

SUMMARY:
A prospective, multi-centric, cohort study to observe the efficacy difference between intensive classic DMARDs and Infliximab(IFX) with methotrexate(MTX) treatment in sever rheumatoid arthritis(RA) 28 joints disease activity score>5.1(DAS28>5.1) patients with poor prognostic factors.Primary objective is compare the difference of clinical remission rate between classic DMARDs and Infliximab with MTX treatment in severe RA patients with poor prognostic factors at week 30.

DETAILED DESCRIPTION:
Primary objective is compare the difference of clinical remission rate between classic conventional disease-modifying antirheumatic drugs(DMARDs) and Infliximab with methotrexate(MTX) treatment in severe RA patients with poor prognostic factors at week 30.

Secondary objectives are compare the differences of laboratory measurements, clinical remission rate, function score and imageological evaluation between classic DMARDs and Infliximab with MTX treatment in severe RA patients with poor prognostic factors at week 14, 30, 54 and 102.

Infliximab arm：Infliximab with MTX treatment: Infliximab 3mg/kg at week 0, 2, 6 and then once every 8 weeks, MTX>7.5mg per week. To observe the results at week 14, 30, 54 and 102 after 6 times IFX treatment. It recommended that continue to receiving IFX treatment after remission for a period of time in good economic condition patients while receiving MTX with hydroxychloroquine(HCQ) or leflunomide(LEF) in poor economic condition patients.

Classic DMARDs treatment arm： Classic DMARDs treatment combination of 2 or 3 drugs, 2-drugs combination is MTX with LEF or Thunder God Vine, 3-drugs combination is MTX with HCQ and LEF or Thunder God Vine for total 30 weeks.

Effective dose: MTX: 10-15mg per week; LEF: 20mg per day; HCQ: 200-400 mg per day; Thunder God Vine: 40-60 mg per day; It recommended that the maintain regimen is MTX with HCQ or LEF after remission for a period of time.

Study is divided into three stages First stage: day -7 to 0

1. Sign informed consent;
2. Examine and verify the inclusion and exclusion criteria;
3. Collect the data of demographic characteristics, history of present illness, signs and symptoms, history of previous illness and concomitant medicine, personal history, allergic history, injury and surgery history;
4. Data of laboratory examinations: Rheumatoid Factor(RF),anti citrullinated protein antibodies(ACPA) ;
5. Safety data: vital signs, blood routine examination, biochemical test;
6. Efficacy data: Erythrocyte Sedimentation Rate(ESR), C Reactive Protein(CRP), 28 joints disease activity score(DAS28 score), Simplified disease activity index(SDAI) score, American College Of Rheumatology(ACR)/European League Against Rheumatism(EULAR) remission ,Sharp van der Heijde scoring(SHARP) score, Magnetic Resonance Imaging(MRI) score, Health Assessment Questionnaire(HAQ) score;

Second stage: week 0 to week 30, follow-up duration I The subjects are randomized assigned to achieve experimental or control treatment for 30 weeks and follow up at week 2, 6, 14, 22 and 30.

1. The follow up items are same at week 2 and week 22: signs and symptoms, ESR, CRP;
2. The follow up items at week 6: signs and symptoms, blood routine examinations, biochemical test, ESR, CRP;
3. The follow up items at week 14: signs and symptoms, ESR, CRP, DAS28 score, SDAI score, ACR/EULAR remission, SHARP score, MRI score, HAQ score;
4. The follow up items at week 30: signs and symptoms, RF, ACPA, blood routine examinations, biochemical test, ESR, CRP, DAS28 score, SDAI score, ACR/EULAR remission, SHARP score, MRI score, HAQ score.

Third stage: Week 30 to 102, follow-up duration II After 30 weeks treatment the subjects are into 72 weeks follow-up duration, the follow up will be conducted at week 38, 46, 54 and 102.

1. The follow up items are same at week 38 and 46: signs and symptoms, ESR, CRP;
2. The follow up items: signs and symptoms, blood routine examinations, biochemical test, ESR, CRP, DAS28 score, ACR/EULAR remission, SHARP score, MRI score, HAQ score;
3. The follow up items at week 102: signs and symptoms, RF, ACPA, blood routine examinations, biochemical test, ESR, CRP, DAS28 score, SDAI score, ACR/EULAR remission, SHARP score, MRI score, HAQ score.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide written informed consent and to comply with the study protocol
2. Age is from 18 to 70 years old
3. To accord with the diagnostic criteria of ACR/EULAR 2010 and the course of disease is less than 2 years;
4. Active RA, DAS28 score is above 5.1
5. At least has one poor prognostic factor including:(1)functional limitations,(2)extra-articular manifestation,(3)positive RF or Anti-Cyclic Citrullinated Peptide(CCP) antibody ,(4)X- ray confirmed bone erosion.

Exclusion Criteria:

1. Received Infliximab or other biologics treatment previously;
2. Abnormal liver function, the level of alanine aminotransferase(ALT) and aspartate amino transferase(AST) is higher than 3 times of upper limit of normal (ULN);
3. Renal dysfunction, the level of serum creatinine is higher than 1.5 times of ULN;
4. Receive live virus or bacterial vaccination currently or 4 weeks before recruitment into the study;
5. Previously affected by tuberculosis or with positive tuberculin test result;
6. Has history of lymphoproliferative disease such as lymphoma or suspected lymphoproliferative disease through signs and symptoms such as lymphadenectasis in posterior cervical triangle, interclavicular or supratrochlear, or splenomegaly (more than 2 cm below the ribs);
7. History of multiple sclerosis or other demyelinating diseases of central nervous system;
8. Be allergic to experimental drug or with serious allergic constitution;
9. Malignancies excluding cured skin basal cell carcinoma or carcinoma in situ of cervix;
10. Systemic active infection, HIV infection or active Hepatitis B or Hepatitis B virus carriers;
11. With serious medical diseases such as cardiac insufficiency (), myocardial ischemia, serious arrhythmia, renal insufficiency, serious liver dysfunction, significant hematological system diseases, hypercortisolism, uncontrollable hypertension and diabetes mellitus;

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2013-08; Primary Completion 2015-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
The rate of subjects achieving DAS<2.6 | at week 30
  The rate of subjects achieving DAS<2.6 at week 30

SECONDARY OUTCOMES:
The rate of subjects achieving DAS<2.6 | at week 14, 54 and 102
  The rate of subjects achieving DAS<2.6 at week 14, 54 and 102
The rate of subjects achieving SDAI<3.3 | at week 14, 30, 54 and 102
  The rate of subjects achieving SDAI<3.3 at week 14, 30, 54 and 102;
The rate of subjects achieving ACR/EULAR remission | at week 14, 30, 54 and 102
  The rate of subjects achieving ACR/EULAR remission at week 14, 30, 54 and 102;
MRI score | at week 14, 30, 54 and 102
  MRI score at week 14, 30, 54 and 102;
The HAQ score | at week 14, 30, 54 and 102
  The HAQ score at week 14, 30, 54 and 102;
The SHARP score | at week 14, 30, 54 and 102
  The SHARP score at week 14, 30, 54 and 102
The level of ESR | at week 2, 6, 14, 22, 30, 54 and 102
  The level of ESR at week 2, 6, 14, 22, 30, 54 and 102
The level of CRP | at week 2, 6, 14, 22, 30, 54 and 102
  The level of CRP at week 2, 6, 14, 22, 30, 54 and 102

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Zhang, Ph.D, Principal Investigator — Director
Locations (3):
- China (3):
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - XIJING Hospital, Xi’an, Shanxi
  - Tianjin medical university general hospital, Tianjin, Tianjin Municipality